CLINICAL TRIAL: NCT00853502
Title: The Effect of Testosterone Replacement on Bone Mineral Density and Bone Microarchitecture in Teenage Boys and Young Adult Men With Anorexia Nervosa
Brief Title: The Effect of Testosterone Replacement on Bone Mineral Density in Boys and Men With Anorexia Nervosa
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Madhusmita Misra, Chief, Pediatric Endocrinology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008P-001902
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Bone Metabolism
Keywords: anorexia nervosa; testosterone; disordered eating; hypogonadism; bone
MeSH Terms: conditions — Anorexia Nervosa; Hypogonadism | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- testosterone cypionate (Active Comparator)
  Interventions: Drug: testosterone cypionate
- bone monitoring (No Intervention)

INTERVENTIONS:
Drug: testosterone cypionate — dose dependent on pubertal stage, intramuscular injection once every 3 weeks for 12 months
  Arms: testosterone cypionate

SUMMARY:
Decreased bone strength is a common and serious medical problem present in many people with anorexia nervosa. Men with anorexia nervosa have lower levels of gonadal steroids such as testosterone. Low testosterone levels have been shown to result in low bone density.

We are investigating whether bone mineral density and bone microarchitecture are abnormal in males with anorexia nervosa and whether supplementation with testosterone would improve both bone mineral density and bone microarchitecture.

DETAILED DESCRIPTION:
Low bone mineral density is a co-morbidity associated with anorexia nervosa that has been shown to persist even after weight gain. Peak bone mass accrual occurs during the adolescent years, and a disruption in this critical process increases the risk for developing persistent deficits in bone density, and possibly increased fracture risk. Multiple variables contribute to the bone mass accrual process in puberty including adequate levels of sex hormones and puberty specific changes in levels of these hormones. Teenage boys with anorexia nervosa have lower bone density than normal weight boys of comparable maturity, and also have decreased levels of testosterone, as well as estradiol, when compared with healthy controls. Although testosterone is an important predictor of bone density in males with anorexia nervosa, the effect of testosterone replacement on bone mass accrual and bone microarchitecture in hypogonadal teenage boys and young adult men with anorexia nervosa is unknown. We hypothesize both bone mass and bone microarchitecture are abnormal in anorexia nervosa and that testosterone replacement in adolescent males with anorexia nervosa will improve both bone mass and microarchitecture.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa
* Teenage boys and young adult men, age 14-30 years
* Hypogonadism indicated by a testosterone level within the lower 25th percentile for pubertal stage or below normal for pubertal stage

Exclusion Criteria:

* Disease or illness known to affect bone metabolism
* Use of medications known to affect bone metabolism, such as corticosteroids or androgenic steroids, within 3 months of study initiation
* Subjects with a z-score less than -2.5 on DXA secondary to concerns of severely low bone mineral density which may require aggressive monitoring

Ages: 14 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
bone metabolism | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Madhusmita Misra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Misra M, Katzman DK, Cord J, Manning SJ, Mendes N, Herzog DB, Miller KK, Klibanski A. Bone metabolism in adolescent boys with anorexia nervosa. J Clin Endocrinol Metab. 2008 Aug;93(8):3029-36. doi: 10.1210/jc.2008-0170. Epub 2008 Jun 10. PMID 18544623